CLINICAL TRIAL: NCT00269750
Title: The Maximum Tolerated Dose and Minimum Effective Dose of OROS® Oxybutynin Compared to Ditropan® (Immediate-release Oxybutynin) in the Treatment of Patients With Urge or Mixed Urinary Incontinence
Brief Title: A Study Comparing the Efficacy and Safety of OROS® Oxybutynin to That of Ditropan® (Immediate-release Oxybutynin) for the Treatment of Patients With Urge or Mixed Urinary Incontinence.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005968
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Urge Incontinence
Keywords: Ditropan®; OROS®; urge; oxybutynin; mixed urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Urge | interventions — oxybutynin

INTERVENTIONS:
Drug: OROS® oxybutynin or Ditropan®

SUMMARY:
The purpose of this study is to compare the efficacy and safety of OROS® oxybutynin to that of Ditropan® (immediate-release oxybutynin) for the treatment of patients with urge or mixed urinary incontinence. Oxybutynin is an antispasmodic, anticholinergic medication for the treatment of the symptoms of overactive bladder.

DETAILED DESCRIPTION:
Ditropan® is indicated for the treatment of urge urinary incontinence, however patients tend to discontinue the medication or decrease the dose due to anticholinergic side effects. OROS® oxybutynin, a continuous release formulation, is expected to have fewer anticholinergic side effects than Ditropan® and may provide equal or better efficacy compared to Ditropan®. This is a randomized, multi-center, double-blind, parallel group, dose-escalation study comparing the efficacy and safety of OROS® oxybutynin to Ditropan® for the treatment of urge or mixed urinary incontinence at the minimum effective dose (MED), the maximum tolerated dose (MTD), or the maximum allowable dose (MAD) permitted under this protocol. Patients in both treatment groups begin study drug treatment at an oxybutynin dose of 5 mg per day. The dose is changed in 5 mg increments at 4- to 7-day intervals, depending on the safety and efficacy of the current dose. The maximum allowable dose for Ditropan® is 20 mg per day, which is the maximum daily adult dose specified in its labeling. Because controlled delivery of oxybutynin by an OROS® dosage form could potentially reduce side effects, it is believed that the drug could possibly be tolerated at doses higher than 20 mg per day. Consequently, the maximum allowable dose for OROS® oxybutynin is 30 mg per day, administered as a single daily dose. The primary measures of effectiveness include the change from baseline in the following assessments: the number of urge urinary incontinence episodes per week, the total number of urinary incontinence episodes, and total void frequency (normal and incontinent). Safety evaluations include the incidence of adverse events, physical examination and medical history, clinical laboratory tests, urinalysis, electrocardiograms (ECGs), vital signs, and the Anticholinergic Effects Assessment (ACEA) questionnaire.

OROS® (oxybutynin chloride) 5 mg tablets, one to six tablets per day (5 mg/day to 30 mg/day) as a single morning oral dose for 11 days up to 70 days, and Ditropan (oxybutynin chloride) 5 mg tablets, one to four tablets per day orally (5 mg per day to 5 mg four times per day) for 10 daysup to 61 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with urge or mixed urinary incontinence, provided that stress urinary incontinence is not the predominant manifestation of mixed urinary incontinence
* Patients who are currently taking immediate release oxybutynin (Ditropan®) hyoscyamine (Levsin®) or propantheline (Pro-banthine®), or who have taken Ditropan in the past for urge or mixed UI. (Patients who have taken Ditropan for urge or mixed urinary incontinence, but who have discontinued the medication should have discontinued due to anticholinergic effects and not due to failure of efficacy)
* Patients who are able to differentiate incontinent episodes associated with urgency from incontinent episodes not associated with urgency when recording incontinent episodes in the diary, who have at least six urge urinary incontinence episodes per week recorded on the Run-in Diary after washout of anticholinergic medications, and who demonstrate that the number of urge incontinent episodes per week is greater than the number of incontinent episodes not associated with urgency per week
* Patients who are in good general health prior to study participation, having normal blood pressure with or without hypertension medication
* Agreeing that a medically acceptable and effective birth control method will be used by the patient and partner throughout the study and for one week following the end of the study

Exclusion Criteria:

* Patients with known treatable genitourinary conditions that may cause incontinence (e.g., urinary tract infection, prostatitis, urinary tract obstruction, bladder tumor, bladder stone, prostate cancer)
* Patients with glaucoma or untreated narrow anterior chamber angles, obstructive bowel disease or severe narrowing of the gastrointestinal tract, obstructive uropathy, or myasthenia gravis
* Patients with known allergy or hypersensitivity to oxybutynin or clinically significant medical problems or other organ abnormality or pathology for whom, administration of oxybutynin would present undue risk
* Male patients with a PSA > 10 ng/mL or a PSA between 4 ng/mL and 10 ng/mL who in the opinion of the investigator require further evaluation or treatment for prostate cancer, or male patients who have had prostate surgery less than nine months before study enrollment. (Prostate pathology from surgery must be benign)
* Patients whose estimated creatinine clearance is less than 50 mL/min or a have hemoglobin level less than 10 g/dL

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 1996-07; Study Completion 1997-02

PRIMARY OUTCOMES:
Change from baseline in: the number of urge urinary incontinence episodes per week; total number of urinary incontinence episodes; total void frequency (normal and incontinent)

SECONDARY OUTCOMES:
Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — Alza Corporation, DE, USA

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- See also: The maximum tolerated dose and minimum effective dose of OROS® oxybutynin compared to Ditropan® in the treatment of patients with urge or mixed urinary incontinence (UI) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=97&filename=CR005968_CSR.pdf